CLINICAL TRIAL: NCT04722809
Title: Efficacy of Botulinum Toxin A in the Treatment of Bruxism-related Symptomatology
Acronym: Botox
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties in recruiting patients, compounded by problems extracting data from the device used in the study.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWETYENGA CRBFC 2020
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Bruxism
MeSH Terms: conditions — Bruxism | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptomatic patients in the context of bruxism (Experimental)
  Interventions: Drug: Botulinum toxin injection; Other: QOL-Brux; Other: Muscular strength of the jaw; Other: Intensity and frequency of episodes of nocturnal bruxism; Other: visual analogue pain scale; Other: Endobuccal and linea alba photographs

INTERVENTIONS:
Drug: Botulinum toxin injection — Injection in the temporal and masseter muscles: in 3 points in the masseter muscles and in 2 points in the temporal muscles.
Other: QOL-Brux — Questionnaire evaluating the symptoms of bruxism Inclusion and 3 months post-injection
Other: Muscular strength of the jaw — Measurement in the jaw with a dynamometer connected to a sensor placed on the 1st molar on the right side.
  At inclusion and 1 month post-injection.
Other: Intensity and frequency of episodes of nocturnal bruxism — Measurements via a portable electromyography system, coupled with a heartbeat sensor (Bruxoff®). Measurements performed during normal sleeping conditions at home before injection and 1 month after.
Other: visual analogue pain scale — Evaluation of jaw pain. At inclusion and 3 months post-injection
Other: Endobuccal and linea alba photographs — anonymous endobuccal and linea alba photographs (line on the inner face of the cheeks as the result of chronic friction).
  At inclusion

SUMMARY:
Bruxism is defined as a parafunction that consists of a clenching of the jaw and/or grinding of the teeth. It can occur when an individual is sleeping or awake or it can be mixed.

Most often, it is primary or idiopathic bruxism, however when it is related to a cause it is qualified as secondary.

Primary bruxism is a condition that is not well known to the general public, but I is very widespread (12% of the adult population). In addition, it can alter quality of life, as a result of associated sleep disorders, concentration disorders, daytime fatigue, chronic pain, etc.

The current treatment for this condition is only symptomatic. Currently, one of the most effective treatments is the intramuscular injection of botulinum toxin A in the muscles of mastication. The progressive anticholinergic action results in a reduction of functional signs (dental pain, periodontal pain, temporomandibular joint pain, tension headaches, neck pain) and physical signs (reduction of the mass of the injected muscles, alba linea, tongue scalloping, limitation or stability of dental damage).

However, these clinical data are practically not objectified in daily practice. Objective criteria would make it possible to measure the effectiveness of the treatment, to follow the patient, and to identify the early symptoms in order to prevent a recurrence.

The aim of the prospective study is to concretely measure the strength and electromyographic activity of the muscles of mastication before and after botulinum toxin injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given written consent.
* Patient between 18 and 64 years of age.
* Patient who has never received botulinum toxins
* Symptomatic patient in the context of bruxism in failure to the usual treatments (analgesic, physiotherapy, relaxation technique and maxillary retainer)
* Woman of childbearing age using an effective method of contraception
* Symptomatic patients in the context of bruxism, without a maxillary disocclusion retainer.

Exclusion Criteria:

* Protected Adult
* Patient not affiliated to the national health insurance system
* Pregnant or breastfeeding woman
* Refusal to take part in the study
* Neuromuscular diseases, including Myasthenia gravis, Myopathies, Amyotrophic Lateral Sclerosis. Lambert-Eaton Syndrome, patients with peripheral motor neuropathies, patients with underlying neurological disorders.
* Patients with a history of cardiovascular disease
* Patients with epilepsy or a previous seizure episode
* Neurogenic impairment of the face (including facial paralysis, polyradiculoneuritis)
* History of dysphagia or pulmonary aspiration
* Injection site infection (masseter and temporal)
* Hypersensitivity or allergy to botulinum toxin or any of its excipients.
* Treatment with aminoglycosides or anticholinesterase agents.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
number of episodes of nocturnal bruxism | 1 month after treatment by botulinum toxin injection
  measurement of the number of bruxism episodes via a portable electromyogram we expect a significant improvement in the number of nocturnal bruxism episodes (decrease in relation to time 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France